CLINICAL TRIAL: NCT05814978
Title: Effects of Scapular Therapeutic Exercise on Essential Biomechanical and Neurophysiological Parameters in Shoulder Pain Conditions With Scapular Impairments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Polytechnic Institute of Porto (Other)
Collaborators: School of Health of Polytechnic Institute of Porto (Unknown); Center for Rehabilitation Research - Human Movement System (Re)habilitation Area (Unknown); Universidade do Porto (Other); Porto Biomechanics Laboratory (Unknown); Center for Interdisciplinary Applied Research in Health, Health School of the Setubal, Polytechnic Institute (Unknown)
Responsible Party: Principal Investigator, Ana Melo, Principal Investigator - PhD grant student, Polytechnic Institute of Porto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CE0108C; SFRH/BD/140874/2018 (Other Grant/Funding Number: Fundação para a Ciência e Tecnologia (FCT), Portugal); UIDB/05210/2020 (Other Grant/Funding Number: Fundação para a Ciência e Tecnologia (FCT), Portugal and the European Union (EU))
Record Dates: First submitted 2023-03-17; First posted 2023-04-18 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Shoulder Pain
Keywords: Shoulder pain; Scapular muscles; Scapular kinematics; Therapeutic exercise
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Scapular Therapeutic Exercise Group (Experimental): Patients in this group will perform therapeutic exercises, recommended for subjects with shoulder pain and focusing the neuromuscular control, stretching and/or strengthening of the scapular muscles
  Interventions: Other: Experimental Scapular Therapeutic Exercise Group

INTERVENTIONS:
Other: Experimental Scapular Therapeutic Exercise Group — All subjects will perform a program of scapular therapeutic exercises including: neuromuscular control/strength - scapular therapeutic exercises that leads to, at least, moderate muscular activity levels; and stretching exercises.
  The intervention period will be of 8 weeks, considering in-person and/or home sessions.

SUMMARY:
Shoulder pain is a prevalent and recurrent condition. After a period of shoulder pain, some adaptations could be found, as in scapular muscles and kinematics and/or in nervous system.

It seems important to assess several biomechanical and neurophysiological outcomes to better characterize shoulder pain conditions and to program an intervention plane.

Therapeutic exercise is one of the treatments used for shoulder pain, however there are still doubts and controversial findings regarding exercise focusing the scapular musculature. Thus, the present study aims to assess the effects of an intervention protocol based on scapular therapeutic exercise.

DETAILED DESCRIPTION:
The study only started after approval of the protocol

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years old
* Chronic (more than 3 months), continuously or intermittently, non-specific or associated with a diagnostic (except if mentioned in the exclusion criteria) shoulder pain of, at least, moderate intensity
* Presenting scapular alterations as scapular dyskinesis (identified at rest or during motion)

Exclusion Criteria:

* History of shoulder fracture, dislocation, tears, infection or neoplasm
* Shoulder surgery
* Cervical and/or thoracic pathologies or pain associated with active movements of these regions
* Neurological disease
* Body mass index out of the range 18,5-30 kg/m2 and muscular skinfold higher than 20mm
* Inability to perform the exercises
* Current practice of competitive/high-level exercise/sport focusing the upper limb

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-04-20 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Change in shoulder pain | Baseline and one week after intervention
  The intensity of pain will be measured with a self-reported 11-point scale (Numerical Rating Pain Scale), with scores ranging from 0 (no pain) to 10 (maximum pain)
Change in shoulder function | Baseline and one week after intervention
  Shoulder functional status will be measured with a self-reported 13 items scale (SPADI), which ranges from 0 (fully functional) to 100 (maximum degree of disability).
Change in scapular muscles activity levels | Baseline and one week after intervention
  Scapular muscles activity levels, during shoulder analytical movements and during a functional task, will be recorded superficially by a wireless electromyographic signal detector system
Change in scapular muscles ratio | Baseline and one week after intervention
  Ratio between scapular muscles activity levels, during shoulder analytical movements and during a functional task, will be calculated considered the superficially eletromyographic data measured by a wireless electromyographic signal detector system.
Change in kinematics | Baseline and one week after intervention
  Scapular kinematics and scapulohumeral rhythm, during shoulder analytical movements and during a functional task, will be measured by inertial sensors and described in degrees (°)
Change in movement quality through time variables | Baseline and one week after intervention
  Movement quality will be assessed considering time to peak acceleration and task completion time, calculated according to the data recorded with inertial sensors
Change in movement quality through trunk compensation | Baseline and one week after intervention
  Movement quality will be also assessed considering the trunk motion, calculated according to the data recorded with inertial sensors
Change in movement quality through smoothness | Baseline and one week after intervention
  Smoothness will be calculated by jerk logarithm of data recorded with inertial sensors

SECONDARY OUTCOMES:
Change in muscle stiffness | Baseline and one week after intervention
  Scapular muscles stiffness will be assessed by myotonometry (using a digital palpation device)
Change in pressure pain threshold | Baseline and one week after intervention
  An assessment point in the shoulder area will be assessed by the application of a mechanical pressure by an algometer
Change in pain-related fear | Baseline and one week after intervention
  Assessed with self-reported scales - Tampa Scale for Kinesiophobia, which ranges from 13 (best) to 52 (worst)
Change in pain catastrophization | Baseline and one week after intervention
  Assessed with a self-reported scale - Pain Catastrophizing Scale, which ranges from 0 (better) to 52 (worst)
Self-impression of change | One week after intervention
  The patient's individual perspective about his/her condition and changes felt considering the intervention received will be assessed by a self-reported scale - Patient global impression of change scale, which range from 0 [no change (or condition has got worse)] to 7 (a great deal better, and a considerable improvement that has made all the difference)

CONTACTS AND LOCATIONS:
Overall Officials: Ana Melo, Principal Investigator — Polytechnic Institute of Porto
Locations (1):
- Center for Rehabilitation Research, School of Health, Polytechnic of Porto, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No